CLINICAL TRIAL: NCT02095769
Title: Pharmacogenomic Testing Of the Elderly To Reduce Morbidity
Acronym: POETRY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Genetics Corporation (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Other Study IDs: 201301
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Genetics of Drug Metabolism
Keywords: Pharmacogenomics; Adverse Drug Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the POETRY Registry is to determine whether data from Pharmacogenomic (PGx) Testing for elderly and disabled patients can help physicians manage patient medication regimens and assess if the testing has an effect on reducing adverse drug events, hospitalizations, and emergency department visits.

The way an individual processes or metabolizes a drug is in part determined by their genes, and there is known to be genetic variation from one human to another. The study of the way in which genes affect an individual's response to drugs is known as "Pharmacogenomics."

ELIGIBILITY:
Inclusion Criteria:

* Subject underwent PGx testing for the alleles appropriate to the target drugs within the prior 90 days ('index PGx test')
* Males and females aged ≥65 years or male and females aged ≥18 years who have a disability
* Subject is able and willing to provide written informed consent
* Subject was receiving at least one medication known to be associated with allelic variation at the time of the index PGx test, including over-the-counter medications
* Subject has a history of at least one target drug-related adverse event (TDAE) over the 12-month period preceding receipt of PGx test results, or has experienced inadequate efficacy from a target drug

Exclusion Criteria:

* Subject is currently hospitalized
* Subject's medical and medication history is unavailable over the 90-day period preceding the receipt of PGx test results
* Subject is unable to provide an accurate history due to mental incapacity
* Subject is known to have undergone prior PGx testing for genes specific to the target drug(s), exclusive of the PGx test relating to this Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 65 and above or subjects aged 18 and above who have a disability will be eligible for inclusion in the study if they are receiving or are planned to receive at least one medication with a metabolic pathway linked to genetic variations ("target drug").
Sampling Method: Non-Probability Sample
Enrollment: 280000 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Meaningful Change in Drug Regimen | 90 days
  The primary endpoint of the study is the binary occurrence of meaningful change in drug regimen, defined in each subject when:
  1. A genotype known to affect a drug the subject is taking is identified, and
  2. The subject's treating physician makes at least one target drug regimen change, dose, substitution, or discontinuation.

SECONDARY OUTCOMES:
Binary occurrence of meaningful change in drug regimen, defined at the drug level over the 90-day period following receipt of PGx test results | 90 days
Binary occurrence of meaningful change in drug regimen, defined at the gene level over the 90-day period following receipt of PGx test results | 90 days
Binary occurrence of whether, in the Investigator's opinion, the subject experienced clinical benefit from drug regimen changes made as a result of the PGx test | 90 days
  Clinical benefit refers to improvement in the subject's condition in the Investigator's opinion
Number of changes in a subject's target drugs, tabulated on a per-subject basis by number and percentage of target drugs and total drugs | 90 days
Binary change (yes/no) in the regimen of drugs controlled by genes of interest over the 90-day period preceding PGx testing compared with the change (yes/no) over the 90-day period following receipt of PGx test results | 90 days
Number of target drug-related adverse events over the 90-day period prior to and following PGx testing | 90 days
Emergency department visits over the 90-day periods prior to and following PGx testing | 90 days
Hospitalizations over the 90-day period prior to and following receipt of PGx test results | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bill Massey, PhD, Principal Investigator — Northwestern University
Locations (8):
- United States (7):
  - Core Insitute, Phoenix, Arizona
  - LifeSpan Institute, La Jolla, California
  - The International Heart & Lung Institute Center for Restorative Medicine, Palm Springs, California
  - Research Physicians Network Alliance, Pembroke Pines, Florida
  - Tallahassee Neurological Institute, Tallahassee, Florida
  - Hypertension Institute, Nashville, Tennessee
  - Diagnostic Clinic of Houston, Houston, Texas
- Research & Cardiovascular Corp., Ponce, PR, Puerto Rico